CLINICAL TRIAL: NCT02174796
Title: Hemodynamic Repercussions of the Correction (Surgical and Non Surgical) of Pectus Excavatum-type Thoracic Deformities
Acronym: PECTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A01811-44
Record Dates: First submitted 2014-04-23; First posted 2014-06-26 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Pectus Excavatum
Keywords: Pectus excavatum; cardiac output; transthoracic impedancemetry
MeSH Terms: conditions — Funnel Chest | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical treatment group (Experimental): patients who chose to undergo a surgical correction (Ravitch or Nuss type intervention).
  intervention: surgical correction (Ravitch or Nuss type intervention).
  Interventions: Procedure: surgical treatment
- Orthopedic treatment group (Experimental): patients who chose an orthopedic treatment by vacuum bell. intervention : orthopedic treatment by vacuum bell.
  Interventions: Procedure: orthopedic treatment

INTERVENTIONS:
Procedure: surgical treatment — patients who chose to undergo a surgical correction (Ravitch or Nuss type intervention).
  Arms: Surgical treatment group
Procedure: orthopedic treatment — orthopedic treatment by vacuum bell.
  Arms: Orthopedic treatment group

SUMMARY:
this non-randomized prospective study of 2 longitudinal cohorts (surgical treatment group or orthopedic treatment group), will evaluate the hemodynamic repercussions of the correction (surgical and non surgical) of pectus excavatum-type thoracic deformities by measuring the cardiac output difference before and after intervention, measured by transthoracic impedancemetry, during an exercise stress test

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking treatment of a pectus excavatum
* Haller index > 3.2
* Desire for treatment
* age between 15 and 40 years old

Exclusion Criteria:

* Cognitive impairment
* Pregnancy
* Contraindication to exercise stress test or general anesthesia
* Coagulation disorders

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Cardiac output difference before and after intervention,during an exercise stress test | 4 months before treatment (initial evaluation E1) just before treatment (intermediate evaluation E2) and 4 months after surgical treatment (TC) or orthopedic treatment (TO) of the deformation (final evaluation E3)
  Cardiac output measured by transthoracic impedancemetry, during an exercise stress test

SECONDARY OUTCOMES:
Rest lung function tests | 4 months before treatment (initial evaluation E1) just before treatment (intermediate evaluation E2) and 4 months after surgical treatment (TC) or orthopedic treatment (TO) of the deformation (final evaluation E3)
Exercise functional capacity | 4 months before treatment (initial evaluation E1) just before treatment (intermediate evaluation E2) and 4 months after surgical treatment (TC) or orthopedic treatment (TO) of the deformation (final evaluation E3)
Exercise cardiac output | 4 months before treatment (initial evaluation E1) just before treatment (intermediate evaluation E2) and 4 months after surgical treatment (TC) or orthopedic treatment (TO) of the deformation (final evaluation E3)
  Exercise cardiac output (measured by transthoracic echocardiography)
Quality of life | 4 months before treatment (initial evaluation E1) just before treatment (intermediate evaluation E2) and 4 months after surgical treatment (TC) or orthopedic treatment (TO) of the deformation (final evaluation E3)
  Quality of life SF36
Mean energy expenditure | 4 months before treatment (initial evaluation E1) just before treatment (intermediate evaluation E2) and 4 months after surgical treatment (TC) or orthopedic treatment (TO) of the deformation (final evaluation E3)
  Mean energy expenditure will be evaluated by metabolic and physical activity monitor "armband" during 3 days (Kcal/min)
Evaluation of postoperative neuropathic pain | 4 months before treatment (initial evaluation E1) just before treatment (intermediate evaluation E2) and 4 months after surgical treatment (TC) or orthopedic treatment (TO) of the deformation (final evaluation E3)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Filaire, Pr, Principal Investigator — Centre Jean Perrin, Service de Chirurgie Thoracique
Locations (5):
- France (5):
  - CHU de Clermont-Ferrand, Médecine du sport et d'explorations fonctionnelles, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU G Montpied, Service de Cardiologie et Maladies Vasculaires, Clermont-Ferrand
  - CHU de Saint-Étienne, Hôpital Bellevue, Médecine du Sport et explorations fonctionnelles, Saint-Etienne
  - CHU de St Etienne, Hôpital Nord, Chirurgie thoracique, Saint-Priest-en-Jarez